CLINICAL TRIAL: NCT00269633
Title: Optimizing Light Wavelength for Treatment of Seasonal Affective Disorder
Brief Title: Research Study of Treatment for Winter Depression With Different Colors of Light
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Apollo Health Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080-19000-J11401
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Seasonal Affective Disorder
Keywords: Seasonal Affective Disorder
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red Light Box 657 nm (Placebo Comparator): Red Light Box 657 nm
  Interventions: Device: Red Light Box 657 nm
- Blue Light Box 467 nm (Active Comparator): Blue Light Box 467 nm
  Interventions: Device: Blue Light Box 467 nm

INTERVENTIONS:
Device: Blue Light Box 467 nm — 467 nm Blue LED Light
  Arms: Blue Light Box 467 nm
Device: Red Light Box 657 nm — 657 nm Red LED Light
  Arms: Red Light Box 657 nm

SUMMARY:
The specific aim of this study is to test the hypothesis that light stimuli concentrated around 467 nm will evoke a significantly stronger therapeutic response in SAD patients compared to light stimuli concentrated around 657 nm at an equal photon density.

The secondary objective of this study is to determine the efficacy of different colors and levels of light in order to optimize therapeutic benefit, while also minimizing side effects and maintaining safety of light exposure.

DETAILED DESCRIPTION:
Studies report as many as 1 out of every 5 Americans is affected by mild to severe Seasonal Affective Disorder (SAD, winter depression). Although the exact cause of this condition is unknown, bright light has proven to be an effective therapeutic treatment for many people with SAD. The light sources that have been traditionally used for treatment of SAD produce white light with great variability in the balance of wavelengths that are emitted across the visible spectrum. Although several studies have attempted to test the effectiveness of different wavelengths for treatment of SAD, the devices used in those studies employed broad bandwidths of light. With the technological advancements in light emitting diodes (LEDs) the production of new light therapy equipment with much narrower bandwidths of light is possible. Side effects of exposure to traditional white light therapy for SAD have included hypomanic activation, irritability, headache, eyestrain and nausea. We hypothesize that when the wavelength of light therapy is optimized, it should be feasible to elicit strong therapeutic benefits with lower light intensities and fewer side effects. Previous studies, approved by the Jefferson IRB and successfully completed by our laboratory have shown that some colors of light are more effective in treating SAD than other colors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Seasonal Affective Disorder
* Over 18 years old
* Stable sleeping pattern with a bedtime no later than 1 a.m.

Exclusion Criteria:

* Pregnant women
* Concurrent psychiatric illness that would preclude compliance with the protocol
* active suicidal or homicidal ideation or plan
* variable psychiatric illness (i.e. rapid cycling disorder or severe premenstrual syndrome)
* individuals with substance abuse or dependence who have not been in remission for at least one year
* individuals taking photosensitizing medications
* individuals with macular degeneration or other ocular conditions which might be adversely affected by light
* less then six weeks after onset of psychotherapeutic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George C Brainard, Ph.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glickman G, Byrne B, Pineda C, Hauck WW, Brainard GC. Light therapy for seasonal affective disorder with blue narrow-band light-emitting diodes (LEDs). Biol Psychiatry. 2006 Mar 15;59(6):502-7. doi: 10.1016/j.biopsych.2005.07.006. Epub 2005 Sep 13. PMID 16165105
- [Background] Brainard GC, Sherry D, Skwerer RG, Waxler M, Kelly K, Rosenthal NE. Effects of different wavelengths in seasonal affective disorder. J Affect Disord. 1990 Dec;20(4):209-16. doi: 10.1016/0165-0327(90)90052-a. PMID 2149726
- [Background] Eastman CI, Young MA, Fogg LF, Liu L, Meaden PM. Bright light treatment of winter depression: a placebo-controlled trial. Arch Gen Psychiatry. 1998 Oct;55(10):883-9. doi: 10.1001/archpsyc.55.10.883. PMID 9783558
- [Background] Lee TM, Chan CC, Paterson JG, Janzen HL, Blashko CA. Spectral properties of phototherapy for seasonal affective disorder: a meta-analysis. Acta Psychiatr Scand. 1997 Aug;96(2):117-21. doi: 10.1111/j.1600-0447.1997.tb09915.x. PMID 9272195
- [Background] Lewy AJ, Kern HA, Rosenthal NE, Wehr TA. Bright artificial light treatment of a manic-depressive patient with a seasonal mood cycle. Am J Psychiatry. 1982 Nov;139(11):1496-8. doi: 10.1176/ajp.139.11.1496. No abstract available. PMID 7137404
- [Background] Lewy AJ, Bauer VK, Cutler NL, Sack RL, Ahmed S, Thomas KH, Blood ML, Jackson JM. Morning vs evening light treatment of patients with winter depression. Arch Gen Psychiatry. 1998 Oct;55(10):890-6. doi: 10.1001/archpsyc.55.10.890. PMID 9783559
- [Background] Oren DA, Brainard GC, Johnston SH, Joseph-Vanderpool JR, Sorek E, Rosenthal NE. Treatment of seasonal affective disorder with green light and red light. Am J Psychiatry. 1991 Apr;148(4):509-11. doi: 10.1176/ajp.148.4.509. PMID 2006698
- [Background] Rosenthal NE, Sack DA, Gillin JC, Lewy AJ, Goodwin FK, Davenport Y, Mueller PS, Newsome DA, Wehr TA. Seasonal affective disorder. A description of the syndrome and preliminary findings with light therapy. Arch Gen Psychiatry. 1984 Jan;41(1):72-80. doi: 10.1001/archpsyc.1984.01790120076010. PMID 6581756

RESULTS

PARTICIPANT FLOW:
Groups:
- Red Light Box 657 nm: LED Red Light Box 657 nm
- Blue Light Box 467 nm: LED Blue Light Box 467 nm
Period: Overall Study
Arm/Group | Red Light Box 657 nm | Blue Light Box 467 nm
Started | 4 | 5
Completed | 3 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Red Light Box: 657 nm
  Red Light Box: 657 nm Red LED Light
- Blue Light Box: 467 nm
  Blue Light Box: 467 nm Blue LED Light
- Total: Total of all reporting groups
Arm/Group | Red Light Box | Blue Light Box | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.8) | 39.2 (10.8) | 39.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Structured Interview Guide for the Hamilton Depression Scale - Seasonal Affective Disorder Version (SIGH-SAD); Weekly for Three Weeks
Description: Outcome for Structured Interview Guide for the Hamilton Depression Scale - Seasonal Affective Disorder Version (SIGH-SAD) reported is the average over 3 weeks. Lower values represent less depressive symptoms. Range is 0-53.
Time Frame: Averaged over Three Weeks During Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Red Light Box 657 nm | Blue Light Box 467 nm
Number analyzed (Participants) | 3 | 5
units on a scale | 16.3 (16.9) | 8 (3.6)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Red Light Box: Red Light Box: 657 nm Blue LED Light
Arm/Group | Red Light Box | Blue Light Box
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No